CLINICAL TRIAL: NCT07405567
Title: Ultrasonographic Evaluation of Diaphragm and Accessory Respiratory Muscles During Weaning in ICU Patients With Pneumonia
Brief Title: Ultrasound Evaluation of Respiratory Muscles During Mechanical Ventilation Weaning in ICU Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa Sevket Yilmaz Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gürcan Güler, Principal Investigator, Bursa Sevket Yilmaz Training and Research Hospital
Other Study IDs: 2024-TBEK 2026/01-03
Record Dates: First submitted 2026-01-30; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pneumonia; Invasive Mechanical Ventilation; Weaning From Mechanical Ventilation in Care Unit; Respiratory Muscle Dysfunction
Keywords: Mechanical Ventilation Weaning; Respiratory Muscle Ultrasound; Diaphragm Ultrasound; Parasternal Intercostal Muscle; Anterior Scalene Muscle
MeSH Terms: conditions — Pneumonia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pneumonia ICU Patients on Invasive Mechanical Ventilation: This cohort includes adult intensive care unit patients admitted with pneumonia who are receiving invasive mechanical ventilation via endotracheal intubation. All participants will undergo serial bedside ultrasonographic assessments of the diaphragm, parasternal intercostal muscles, and anterior scalene muscles during the weaning process. No therapeutic intervention is assigned as part of the study, and all clinical management decisions, including ventilator settings and weaning strategies, are determined by the treating ICU team according to standard care.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study with no assigned therapeutic intervention. Serial ultrasonographic assessments of respiratory muscles are performed for observational and data collection purposes only, and all clinical care and weaning decisions are made by the treating intensive care unit team according to standard practice.

SUMMARY:
Patients with pneumonia who require invasive mechanical ventilation in the intensive care unit (ICU) often experience difficulties during the process of being separated from the breathing machine (weaning). Failure of weaning is associated with longer ventilation duration, prolonged ICU stay, and increased risk of complications and death. Therefore, simple and reliable bedside tools are needed to better understand respiratory muscle function and to help predict weaning outcomes.

This prospective, observational, single-center study aims to evaluate respiratory muscle function using bedside ultrasound in adult ICU patients with pneumonia receiving invasive mechanical ventilation. The diaphragm, parasternal intercostal muscles, and anterior scalene muscles will be assessed using ultrasound during the weaning process. Measurements will be performed serially, starting from the first day when patients demonstrate meaningful spontaneous breathing effort and continuing until successful extubation, tracheostomy, or ICU mortality.

Ultrasound measurements of muscle thickness and thickening fraction will be analyzed in relation to weaning outcomes. In addition, ventilator parameters and commonly used weaning indices will be recorded at the time of each ultrasound assessment. The findings of this study are expected to improve understanding of respiratory muscle involvement during weaning and may contribute to earlier identification of patients at risk of weaning failure.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational, single-center cohort study conducted in the intensive care unit (ICU). Adult patients (≥18 years) admitted to the ICU with pneumonia and receiving invasive mechanical ventilation via endotracheal intubation will be eligible for inclusion. Patients with known neuromuscular diseases, high cervical spinal cord injury, prior major neck, thoracic, or diaphragmatic surgery, acute thoracic trauma, pneumothorax, central nervous system pathology, or those receiving continuous neuromuscular blockade will be excluded.

Patients will be followed from ICU admission until one of the following outcomes occurs: successful extubation, tracheostomy, or ICU mortality. The first 24 hours after ICU admission will be defined as ICU Day 1. Disease severity and baseline characteristics will be assessed on ICU Day 1 using the APACHE II, SOFA, frailty index, and Charlson Comorbidity Index scores. Sedation level will be evaluated daily using the Richmond Agitation-Sedation Scale (RASS).

The first day on which the patient demonstrates meaningful spontaneous breathing effort, defined as a RASS score of -3 or higher, will be designated as Measurement Day 0. Ultrasonographic assessments of respiratory muscles will be performed daily for the first three days starting from Measurement Day 0 and every 48 hours thereafter until extubation or another study endpoint is reached. Days with deep sedation (RASS -4 or -5) will be recorded, and only structural muscle thickness measurements will be obtained on those days.

All ultrasound measurements will be performed at the bedside in the supine position under standardized conditions. Ventilator settings will be kept unchanged for at least 30 minutes prior to measurements, and no airway suctioning or position changes will occur within 15 minutes before data acquisition. For each parameter, measurements will be averaged over three consecutive respiratory cycles obtained during a stable ventilation period.

Diaphragm assessment will be performed on the right hemidiaphragm using a low-frequency convex probe at the zone of apposition between the 9th and 10th intercostal spaces along the anterior axillary line. End-expiratory diaphragm thickness will be recorded on all measurement days. On days with RASS ≥ -3, end-inspiratory thickness will also be measured, and diaphragm thickening fraction will be calculated.

Parasternal intercostal muscles will be evaluated using a high-frequency linear probe at the right second and third intercostal spaces along the parasternal line. End-expiratory thickness will be measured on all days, and thickening fraction will be calculated on days with adequate spontaneous breathing effort.

Anterior scalene muscle assessment will be performed using a linear probe at the C6 level, positioned deep to the sternocleidomastoid muscle and lateral to the carotid artery. End-expiratory thickness will be measured daily, and thickening fraction will be calculated on days with RASS ≥ -3.

During each ultrasound session, ventilator mode, pressure support (if applicable), positive end-expiratory pressure (PEEP), fraction of inspired oxygen (FiO₂), respiratory rate, tidal volume, minute ventilation, and peripheral oxygen saturation will be recorded simultaneously. When available, indices reflecting respiratory drive and inspiratory muscle strength, including P0.1, negative inspiratory force (NIF), rapid shallow breathing index (RSBI), and the compliance-rate-oxygenation-pressure (CROP) index, will also be documented. Intra-abdominal pressure will be measured using the intravesical technique at predefined time points.

Ultrasonographic respiratory muscle parameters and their temporal changes will be analyzed in relation to weaning outcomes, with the aim of identifying markers associated with weaning failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the intensive care unit with a diagnosis of pneumonia
* Receiving invasive mechanical ventilation via endotracheal intubation
* Expected to undergo a weaning process from mechanical ventilation
* Written informed consent obtained from the patient or legally authorized representative

Exclusion Criteria:

* Known neuromuscular disease affecting respiratory muscles
* High cervical spinal cord injury
* History of major neck, thoracic, or diaphragmatic surgery
* Acute thoracic trauma or pneumothorax
* Central nervous system pathology affecting respiratory drive
* Continuous neuromuscular blocking agent use
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who are admitted to the intensive care unit with pneumonia and require invasive mechanical ventilation via endotracheal intubation. Patients are followed prospectively during the weaning process from mechanical ventilation and undergo serial bedside ultrasonographic assessment of respiratory muscles as part of observational data collection. All patients receive standard intensive care management as determined by the treating clinical team.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Weaning Failure | From Measurement Day 0 until ICU discharge, up to 72 hours after extubation
  Weaning failure is defined as the need for reintubation within 72 hours after planned extubation, requirement for tracheostomy, or death occurring in the intensive care unit before successful liberation from invasive mechanical ventilation.

SECONDARY OUTCOMES:
Diaphragm Thickening Fraction (TFdi) | From the onset of meaningful spontaneous breathing effort (first day with Richmond Agitation-Sedation Scale ≥ -3) until extubation, tracheostomy, or ICU death, assessed up to 28 days.
  Diaphragm thickening fraction calculated from end-expiratory and end-inspiratory diaphragm thickness measurements obtained by bedside ultrasound on days with meaningful spontaneous breathing effort (RASS ≥ -3).
Parasternal Intercostal Muscle Thickening Fraction (TFic) | From the onset of meaningful spontaneous breathing effort (first day with Richmond Agitation-Sedation Scale ≥ -3) until extubation, tracheostomy, or ICU death, assessed up to 28 days.
  Parasternal intercostal muscle thickening fraction measured by ultrasound at the right second and third intercostal spaces on days with adequate spontaneous breathing effort (RASS ≥ -3).
Anterior Scalene Muscle Thickening Fraction (STF) | From the onset of meaningful spontaneous breathing effort (first day with Richmond Agitation-Sedation Scale ≥ -3) until extubation, tracheostomy, or ICU death, assessed up to 28 days.
  Anterior scalene muscle thickening fraction assessed by bedside ultrasound at the C6 level on days with meaningful spontaneous breathing effort (RASS ≥ -3).
Respiratory Drive and Weaning Indices | From the onset of meaningful spontaneous breathing effort (first day with RASS ≥ -3) until the first occurrence of extubation, tracheostomy, or ICU death, whichever occurs first, assessed up to 28 days.
  Commonly used weaning and respiratory drive parameters including P0.1, negative inspiratory force (NIF), rapid shallow breathing index (RSBI), and CROP index recorded concurrently with ultrasound assessments when available.
Ventilator Parameters During Weaning | From the onset of meaningful spontaneous breathing effort (first day with RASS ≥ -3) until the first occurrence of extubation, tracheostomy, or ICU death, whichever occurs first, assessed up to 28 days.
  Ventilator-related parameters including ventilator mode, pressure support, positive end-expiratory pressure (PEEP), fraction of inspired oxygen (FiO₂), respiratory rate, tidal volume, minute ventilation, and peripheral oxygen saturation recorded at the time of each ultrasound evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Principal Investigator, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy considerations and the absence of a predefined data-sharing agreement for this single-center observational study.

REFERENCES:
- [Result] Bhattacharya D, Esquinas AM, Mandal M. Parasternal Intercostal Muscle Thickness Fraction (PICTF%): Ultrasound a New Tool for Weaning Prediction? Indian J Crit Care Med. 2024 Apr;28(4):404. doi: 10.5005/jp-journals-10071-24665. PMID 38585317
- [Result] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624